CLINICAL TRIAL: NCT07220720
Title: Inclusion of POSLUMA® ((18)F-rhPSMA-7.3) PET-CT Imaging Improves Diagnostic Accuracy of Clinically-Significant Prostate Cancer Diagnosis in Men With PIRADS 2 and 3 Lesions on MRI
Brief Title: POSLUMA® (18F-rhPSMA-7.3) PET-CT for PIRADS 2/3 Lesions
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB202401666
Record Dates: First submitted 2025-06-03; First posted 2025-10-24 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-02

CONDITIONS: Prostate
Keywords: prostate cancer; posluma; pirads 2; pirads 3; prostate biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- POSLUMA PET scan (Experimental): Eligible participants will undergo a PSMA PET scan after infusion of POSLUMA imaging agent.
  Interventions: Drug: Flotufolastat F 18

INTERVENTIONS:
Drug: Flotufolastat F 18 — A PSMA-targeted PET imaging agent used to detect and locate prostate cancer during PET scans that will be administered one time to each study subject.
  Other Names: (18)F-rhPSMA-7.3; POSLUMA

SUMMARY:
The goal of this study to determine if using the (18)F-rhPSMA-7.3 PET-CT scan can improve the ability to spot serious prostate cancer in patients who have uncertain MRI results. These uncertain results include MRI results that showed a PIRADS 2 or PIRADS 3 area on the prostate. The investigators want to find out if this new test is better to detect prostate cancer than just doing a biopsy based on MRI alone.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is willing to provide signed informed consent and is able to comply with all required study-related procedures, where safe and feasible.
2. The patient is male and at least 18 years of age.
3. The patient has not previously undergone a prostate biopsy.
4. The patient underwent a pelvic mpMRI within the last 90 days for the detection of potential prostate cancer (Pca).
5. The patient is a candidate for a targeted MRI/US biopsy and is scheduled to undergo the procedure. Only patients scheduled for a biopsy before recruitment will be considered candidates.
6. The patient has PIRADS 2 and/or PIRADS 3 lesions detected by a board-certified radiologist.

Exclusion Criteria:

1. Patients with a prior diagnosis of prostate cancer.
2. Patients with any medical condition or circumstance that, in the investigator's opinion, could compromise the study data or prevent the patient from fulfilling the study requirements.
3. Patients participating in another interventional clinical trial within the past 30 days.
4. Patients with known hypersensitivity to the active substance or any excipients of flotufolastat F 18 PET-CT.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2030-07-15 (Estimated); Study Completion 2032-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in positive predictive value (PPV) | From enrollment to the end of treatment visit at roughly 12 weeks.
  Evaluate the change in PPV for detecting clinically significant prostate cancer (csPCa) cores by comparing results from mpMRI alone (PIRADS 2 and 3 lesions) to the combination of mpMRI with flotufolastat F 18 PET-CT.
Change in negative predictive value (NPV) | From enrollment to the end of treatment visit at roughly 12 weeks.
  Measure the change in NPV for detecting csPCa cores by comparing mpMRI findings alone (PIRADS 2 and 3 lesions) with the combined approach of mpMRI and flotufolastat F 18 PET-CT.
Improvement in Accuracy | From enrollment to the end of treatment visit at roughly 12 weeks
  Assess the improvement in accuracy (accuracy defined as [(true positive + true negative) / total number of subjects] when using the combined imaging approach of flotufolastat F 18 PET-CT with mpMRI versus mpMRI alone in patients with PIRADS 2 and 3 lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- UF Health - Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided